CLINICAL TRIAL: NCT03313232
Title: Low Dose Exposure to Oxidized R-limonene - A Double Blinded Vehicle Controlled Repeated Open Application Test (ROAT) Study
Brief Title: Low Dose Exposure to Oxidized R-limonene - A Repeated Open Application Test (ROAT) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev and Gentofte Hospital (Other)
Collaborators: University of Copenhagen (Other); Sahlgrenska University Hospital (Other); Göteborg University (Other)
Responsible Party: Principal Investigator, Niels Højsager Bennike, Principal investigator, Herlev and Gentofte Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: HGH-2017-017
Record Dates: First submitted 2017-10-03; First posted 2017-10-18 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Allergic Contact Dermatitis Due to Cosmetics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fragrance allergic patients (Experimental): Patients with a previous positive patch test to oxidized R-Limonene. Patients will have an initial patch test dilution series with oxidized R-limonene performed on the back followed by twice daily exposure to oxidized R-limonene at three different concentrations and a vehicle control on the forearms for up to three weeks.
  Interventions: Other: ROAT with oxidized R-limonene at 1%, 0.3% and 0.1%
- Possible fragrance allergic patients (Experimental): Patients with a previous doubtful patch test to oxidized R-limonene. Patients will have an initial patch test dilution series with oxidized R-limonene performed on the back followed by twice daily exposure to oxidized R-limonene at three different concentrations and a vehicle control on the forearms for up to three weeks.
  Interventions: Other: ROAT with oxidized R-limonene at 1%, 0.3% and 0.1%
- Healty controls (Experimental): Healthy controls with no contact allergy to oxidized R-limonene. Healthy controls will have en initial diagnostic patch test with oxidized R-limonene performed followed by twice daily exposure to oxidized R-limonene at one concentration and a vehicle control on the forearms for up to three weeks.
  Interventions: Other: ROAT with oxidized R-limonene at 1%

INTERVENTIONS:
Other: ROAT with oxidized R-limonene at 1%, 0.3% and 0.1% — A twice daily repeated open application test (ROAT) study for up to three weeks of exposure to oxidized R-limonene at 1%, 0.3% and 0.1% concentrations
  Arms: Fragrance allergic patients; Possible fragrance allergic patients
Other: ROAT with oxidized R-limonene at 1% — A twice daily repeated open application test (ROAT) study for up to three weeks of exposure to oxidized R-limonene at a 1% concentration
  Arms: Healty controls

SUMMARY:
This study evaluates the clinical and molecular effect of daily exposure to low doses of the fragrance contact allergen oxidized R-limonene. Three groups of participants are included: 1) Patients with a previous positive patch test to oxidized R-Limonene, 2) patients with a previous doubtful patch test to oxidized R-limonene and 3) healthy controls with no contact allergy to oxidized R-limonene

ELIGIBILITY:
Inclusion Criteria:

* Positive patch test (at least one reading) or doubtful patch test (at least two readings) to oxidized R-limonene 3% pet. (with 0.33% hydroperoxides content) according to international guidelines, within the last five years.
* Aged 18 years or older
* Received written and verbal information on the study.
* Signed written consent form.

Exclusion Criteria:

* Active eczema in test areas.
* Pregnancy or breast feeding.
* Treatment with topical corticosteroids or other immune-suppressants on/near test areas within two weeks prior to study start.
* Systemic immune-suppressant treatment within seven days prior to study start.
* UV exposure of test areas within three weeks prior to study start.
* Unable to cooperate or communicate with the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2018-04-09 (Actual); Study Completion 2018-04-09 (Actual)

PRIMARY OUTCOMES:
Positive ROAT (minimum score of 5) | Day (D) 21
  Proportion (%) of participants with a positive ROAT

SECONDARY OUTCOMES:
Minimal eliciting concentration (MEC) | Day (D) 7
  Threshold concentration for a positive patch test

OTHER OUTCOMES:
Epidermal inflammatory markers | Positive ROAT or Day (D) 21
  Levels of inflammatory markers (e.g. IL-1beta) from tape stripping of ROAT test areas

CONTACTS AND LOCATIONS:
Locations (2):
- Department of Dermatology and Allergy, Gentofte University Hospital, Hellerup, DK, Denmark
- Department of Occupational and Environmental Dermatology, Sahlgrenska University Hospital, Gothenburg, SE, Sweden